CLINICAL TRIAL: NCT00003679
Title: A Randomised Comparative Trial of Adriamycin + Taxotere vs. Adriamycin + Cyclophosphamide as Primary Medical Therapy for Patients With Potentially Operable Breast Cancer Greater Than or Equal to 3 cm Diameter, Locally Advanced, or Inflammatory Disease
Brief Title: Combination Chemotherapy in Treating Women With Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066780; SCTN-BR9809; EU-98053
Record Dates: First submitted 1999-11-01; First posted 2003-12-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether doxorubicin plus docetaxel is more effective than doxorubicin plus cyclophosphamide for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of doxorubicin in combination with either docetaxel or cyclophosphamide in treating women who have previously untreated, advanced, or inflammatory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy (response rate) and toxicity of doxorubicin in combination with either docetaxel or cyclophosphamide as primary therapy regimens in patients with locally advanced or inflammatory breast cancer.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center and operability. Patients are randomized to one of two treatment arms. Arm I: Patients receive docetaxel IV followed by doxorubicin IV once every 3 weeks. Arm II: Patients receive doxorubicin IV and cyclophosphamide IV once every 3 weeks. Patients receive a maximum of 6 courses of treatment in the absence of disease progression and unacceptable toxicity. Patients then undergo surgery (if operable) followed by more chemotherapy (if node positive), radiation therapy, and oral tamoxifen for 5 years (at the discretion of the investigator for estrogen receptor-negative patients). Patients are followed at 12, 18, and 24 months, and then annually for at least 5 years.

PROJECTED ACCRUAL: A total of 350 patients (175 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven previously untreated locally advanced or inflammatory breast cancer Potentially operable disease Tumor at least 3 cm in diameter No metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 60 Sex: Female Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: PT and aPTT normal Bilirubin normal (except in patients with benign congenital hyperbilirubinemia) AST/ALT no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 1.5 times ULN No active hepatitis B or C Liver biopsy normal (if positive serology for hepatitis B or C) Renal: Creatinine normal Cardiovascular: Adequate cardiac function No active cardiac disease Other: Not pregnant Fertile patients must use effective contraception No other serious medical or psychiatric disease No prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No prior therapy for breast cancer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 1998-11

CONTACTS AND LOCATIONS:
Overall Officials: T.R.J. Evans, Study Chair — Beatson Institute for Cancer Research - Glasgow
Locations (1):
- C.R.C. Beatson Laboratories, Glasgow, Scotland, United Kingdom